CLINICAL TRIAL: NCT05114356
Title: Cervical Interbody Fusion Device Patient Registry
Status: Terminated | Type: Observational
Why Stopped: Sponsor decision
Sponsor: Restor3D (Industry)
Responsible Party: Sponsor
Other Study IDs: restor3d-001
Record Dates: First submitted 2021-10-20; First posted 2021-11-10 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Degenerative Disc Disease
MeSH Terms: conditions — Intervertebral Disc Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Study group: Patients being treated for degenerative disc disease
  Interventions: Device: TIDAL Cervical Interbody Fusion implant

INTERVENTIONS:
Device: TIDAL Cervical Interbody Fusion implant — Cervical interbody fusion device

SUMMARY:
The registry has been designed as a prospective, observational program for patients undergoing anterior cervical discectomy and fusion (ACDF) procedures treated with TIDAL cervical interbody fusion device. The ultimate goal of the study is to aid in the development of treatment pathways and improved patient care. All patients who agree to participate in the registry will sign an informed consent form and subsequently be treated by their surgeon with the device in either an inpatient or outpatient facility.

DETAILED DESCRIPTION:
The registry is design to collect data prospectively on patients undergoing spinal fusion using the TIDAL cervical interbody fusion device. Patients will be enrolled in the registry after reviewing the protocol with their health care provider and signing the informed consent. Data will be collected at recommended time points based on the standards of care of the participating sites. The registry will serve as a database in which retrospective analysis and exploratory analysis of specific research questions will be answered.

Follow up visits will be defined by the treating physicians based on their standard practice. Typical clinical follow up schedules for patients undergoing this type of surgery are pre-operative and 12 months post-operative.

ELIGIBILITY:
Inclusion Criteria:

* Neck and arm pain for a minimum of 6 weeks before surgery that is recalcitrant to nonoperative treatment modalities, such as physical therapy, reduced activities, and anti-inflammatory medications.
* Radiographic evidence of cervical disc disease that is documented on dynamic radiographs and magnetic resonance imaging (MRI).

Exclusion Criteria:

* Medical condition that required medication, such as steroids or nonsteroidal anti-inflammatory medications, that could interfere with fusion.

There are no restrictions on sex or ethnicity.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with degenerative disc disease of the cervical spine, and being surgically treated for degenerative cervical disc disease using a 3D printed titanium interbody cage
Sampling Method: Non-Probability Sample
Enrollment: 73 (Actual)
Dates: Start 2021-11-08 (Actual); Primary Completion 2024-05-22 (Actual); Study Completion 2024-05-22 (Actual)

PRIMARY OUTCOMES:
Change in Oswestry Disability Index (ODI)/Neck Disability Index (NDI) Score Range 0-50 at 1 year post-operative from a pre-operative baseline | 1 year
  ODI/NDI Score Range: 0-50 0-4 No disability 5-14 Mild disability 15-24 Moderate disability 25-34 Severe disability >34 Complete disability
Change in VAS Pain at 1 year post-operative from a pre-operative baseline | 1 year
  VAS PAIN SEVERITY SCALE ranges from 0-10. A score of zero (0) means 'no pain' and a ten (10) means 'worst imaginable pain'

SECONDARY OUTCOMES:
Improvement in patient reported short-form 36 (SF36) scores at 1 year post-operative from a pre-operative baseline | 1 year
  Questionnaire of generic, coherent, and easily administered quality-of-life measures.
Rate of Successful Fusion Based on Radiological Assessment at 1 Year Post-op | 1 year
  Assessment of fusion

CONTACTS AND LOCATIONS:
Locations (1):
- Orthopaedic Institute of Western Kentucky, Paducah, Kentucky, United States